CLINICAL TRIAL: NCT02879695
Title: A Phase 1 Study of Blinatumomab in Combination With Checkpoint Inhibitor(s) of PD-1 (Nivolumab) or Both PD-1 (Nivolumab) and CTLA-4 (Ipilimumab) in Patients With Poor-Risk, Relapsed or Refractory CD19+ Precursor B-Lymphoblastic Leukemia
Brief Title: Blinatumomab and Nivolumab With or Without Ipilimumab in Treating Patients With Poor-Risk Relapsed or Refractory CD19+ Precursor B-Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01300; NCI-2016-01300 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ETCTN10030; 10030 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10030 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Results first posted 2024-10-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Recurrent B Acute Lymphoblastic Leukemia; Recurrent Mixed Phenotype Acute Leukemia; Refractory B Acute Lymphoblastic Leukemia; Refractory Mixed Phenotype Acute Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia, Biphenotypic, Acute | interventions — Specimen Handling; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Biopsy; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (blinatumomab, nivolumab, ipilimumab) (Experimental): Patients receive blinatumomab IV continuously on days 1-28. Treatment repeats every 42 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive nivolumab IV over 30 minutes on day 11 and then every 2 weeks for up to year. Some patients also receive ipilimumab IV over 90 minutes on day 11 and then every 6 weeks for up to 1 year. Patients also undergo bone marrow aspiration and biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration and Biopsy; Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase I trial studies the side effects and best dose of blinatumomab when given with nivolumab alone or nivolumab and ipilimumab in treating patients with poor-risk CD19+ precursor B-lymphoblastic leukemia that has come back after a period of improvement (relapsed) or has not responded to treatment (refractory). Immunotherapy with monoclonal antibodies, such as blinatumomab, nivolumab, and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of the blinatumomab given in combination with nivolumab alone, or in combination with both nivolumab and ipilimumab in subjects with poor-risk, relapsed or refractory CD19+ pre-B cell acute lymphoblastic leukemia (ALL) or CD19+ mixed phenotype acute leukemia (MPAL).

II. To determine the maximum tolerated dose (MTD) of the combination of blinatumomab plus nivolumab, and blinatumomab plus both nivolumab and ipilimumab and to further confirm the safety of the combination therapy in subjects with poor-risk, relapsed or refractory CD19+ pre-B cell ALL or CD19+ mixed phenotype acute leukemia (MPAL).

SECONDARY OBJECTIVES:

I. To observe and record anti-leukemia activity of blinatumomab and nivolumab, and blinatumomab plus both nivolumab and ipilimumab, including the effects on minimal residual disease (MRD).

II. To assess preliminary anti-leukemia activity in expansion cohorts of patients with poor-risk, relapsed or refractory CD19+ precursor B-lymphoblastic leukemia, or CD19+ mixed phenotype acute leukemia (MPAL).

EXPLORATORY OBJECTIVES:

I. To examine changes in absolute lymphocyte count and distribution of T cell subsets (CD4+, CD8+, regulatory T cells [Tregs], effector T cells [Teffs]) and their differentiation status, natural killer (NK) cells, and B cells before and post-blinatumomab, and immune checkpoint inhibitor(s) therapy in both peripheral blood and the bone marrow microenvironment.

II. To explore changes in T cell co-signaling receptors expression in defined T cell subpopulations and their canonic transcription factor expression in both peripheral blood and bone marrow before and post-blinatumomab, and immune checkpoint inhibitor(s) therapy.

III. To examine changes in expression of co-signaling molecules on leukemia blasts (CD10+/CD19+/CD34+) before and after treatment with blinatumomab and checkpoint inhibitors.

IV. To examine the serum levels of cytokines before and after treatment with blinatumomab and checkpoint inhibitors, including the levels of sCTLA-4.

V. To perform immune profiling of T cell repertoire and characterize T cell transcriptional signature before and after treatment.

OUTLINE: This is a safety and tolerability study of blinatumomab given in combination with nivolumab alone, or in combination with both nivolumab and ipilimumab.

Patients receive blinatumomab intravenously (IV) continuously on days 1-28. Treatment repeats every 42 days for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive nivolumab IV over 30 minutes on day 11 and then every 2 weeks for up to year. Some patients also receive ipilimumab IV over 90 minutes on day 11 and then every 6 weeks for up to 1 year. Patients also undergo bone marrow aspiration and biopsy and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY CRITERIA
* Patients must have suspected refractory or relapsed pre-B cell ALL or mixed phenotype acute leukemia (MPAL), or if newly diagnosed, the patient must be 60 years of age or older
* Bone marrow and/or peripheral blood specimens will be submitted for correlative studies; patients who have a dry tap will still be eligible
* REGISTRATION ELIGIBILITY CRITERIA
* Patients must have histologically or cytologically confirmed by the local institution CD19+ precursor B-acute lymphoblastic leukemia (pre-B cell ALL) OR CD19+ mixed phenotype acute leukemia (MPAL): a) with relapse following or refractory to at least one prior line of therapy if older than 21 years; b) in second or higher relapse or refractory to at least two prior lines of therapy if 21 years old and younger (16-21); c) or they must have a new diagnosis of pre-B cell ALL or CD19+ MPAL but are >= 60 years old and are either not a candidate for or do not wish to receive traditional induction chemotherapy
* The evidence of CD19+ expression on leukemia cells must be confirmed by pathology review of the bone marrow and/or peripheral blood specimens (flow cytometry and/or immunohistochemistry) collected at the time of current relapse and prior to the initiation of therapy
* Patients with Philadelphia chromosome (Ph) positive (+) pre-B cell ALL OR Ph+ MPAL will be eligible if they have been refractory to or intolerant of treatment with at least 1 second-generation or third-generation tyrosine kinase inhibitor (TKI)
* Patients who were treated with blinatumomab in the past will be allowed on the study as long as they have persistent CD19 expression on leukemia cells and did not experience unacceptable toxicities with prior blinatumomab administration; patients who were treated with chimeric antigen receptor (CAR)-modified T cells targeting CD19 in the past will be allowed on the study as long as they have persistent CD19 expression on leukemia cells
* Patients with a history of allogeneic hematopoietic stem cell transplantation (HSCT) will be eligible if they are more than 90 days removed from the date of stem cell infusion, have no evidence of acute graft-versus-host disease (GVHD) or active chronic (grade 2-4) GVHD, and are off of all transplant-related immunosuppression for at least 2 weeks
* Age >= 16 years. Because no dosing or adverse event data are currently available on the use of blinatumomab in combination with nivolumab ± ipilimumab in pediatric patients, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG)/Karnofsky performance status of 0-2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Total bilirubin =< 2.0 mg/dL (except patients with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x upper limit of normal (ULN)
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula)
* The effects of nivolumab, ipilimumab, and blinatumomab on the developing human fetus are unknown; for this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP should use an adequate method to avoid pregnancy for 23 weeks after the last dose of investigational drug; women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of treatment on the study; women must not be breastfeeding; men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab +/- ipilimumab and blinatumomab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception

  * Note: Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately
* Adequate pulmonary function as assessed by oxygen saturation >= 90% when ambulating and not requiring supplemental oxygen
* Patients with a known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) will be eligible if:

  * They are generally healthy from an HIV perspective and on a stable anti-retroviral regimen for > 6 months
  * They have had no AIDS-defining conditions in the past 12 months other than historically low CD4+ cell counts
  * They have an undetectable viral load on standard assays
* Patients with a known history of hepatitis C (HCV) will be eligible if they have an undetectable viral load; if the patient received treatment for HCV, then that treatment must have been completed at least three weeks prior to enrollment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or other systemic therapy or radiotherapy, or those who have not recovered from adverse events due to prior administered agents as follows: chemotherapy, radiotherapy or surgery =< 3 weeks prior to entering the study, targeted therapy (e.g., TKI) =< 1 week prior to entering the study; autologous HSCT =< 6 weeks prior to entering the study; investigational drug or immunotherapy (e.g. rituximab) =< 4 weeks prior to entering the study; prophylactic intrathecal chemotherapy within one week of enrollment allowed; patients will be allowed to receive cytoreduction with hydroxyurea, 6-mercaptopurine, corticosteroids (dexamethasone, prednisone or similar) or cyclophosphamide provided that it is discontinued at least 24 hours prior to the initiation of study treatment; pre-phase treatment with dexamethasone 10 mg/m^2 (maximum total 24 mg per day) for up to 5 days is required for patients with bone marrow blasts more than 50%, peripheral blood blasts of 15,000/uL or higher, or elevated lactate dehydrogenase suggesting rapidly progressing disease as per investigator's assessment; pre-phase treatment must be stopped at least 24 hours prior to the initiation of blinatumomab
* Patients who are receiving any other investigational agents
* Patients should be excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Patients with active central nervous system leukemia are excluded from this clinical trial because they may develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; patients with a history of central nervous system (CNS) leukemia but no active disease at the time of enrollment are eligible; the absence of CNS disease must be confirmed by flow cytometric and cytologic examination of the cerebrospinal fluid (CSF) within 7 days of study enrollment
* Active leukemia in the testes or isolated extramedullary relapse; patients with a history of treated leukemia in testes but no active disease at the time of enrollment are eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, ipilimumab, or blinatumomab
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, active, uncontrolled infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements; patients with infection under treatment and controlled with antibiotics are eligible
* Pregnant women are excluded from this study because nivolumab and ipilimumab have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab and ipilimumab, breastfeeding should be discontinued if the mother is treated with nivolumab and ipilimumab; these potential risks may also apply to blinatumomab
* History of any chronic hepatitis including alcoholic, non-alcoholic steatohepatitis (NASH), drug related, autoimmune, chronic viral positive tests for hepatitis B virus surface antigen (HBsAg), hepatitis B core antibody (anti-HBc) in the absence of hepatitis B surface antibody (anti-HBs), or a positive hepatitis C (HCV) viral load; these patients are excluded due to the risk for autoimmune hepatitis with immune checkpoint inhibitors exacerbating their known liver disease as well as the unknown risk for hepatitis B and/or C reactivation with blinatumomab and immune checkpoint inhibitors
* Subjects with active autoimmune disease, a history of known or suspected autoimmune disease or a history of a syndrome requiring systemic corticosteroids (> 10 mg daily of prednisone equivalent) except for the treatment of malignancy with the exception of:

  * Isolated vitiligo
  * Resolved childhood atopy
  * History of a positive antinuclear antibody (ANA) titer without associated symptoms or history of symptoms of an autoimmune disorder
  * Controlled thyroid disorders
  * Type I diabetes mellitus
  * Psoriasis, Sjogren's syndrome, and arthropathies not requiring systemic treatment
  * Autoimmune diseases: these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, autoimmune vasculitis, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen), or as pre-phase treatment for cytoreduction; patients will receive steroids with blinatumomab to reduce cytokine release syndrome (CRS) as specified in the protocol
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study
* Patients who have a history of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, psychosis, or other significant CNS abnormalities; a history of treated CNS leukemia will be allowed if recent CNS studies confirm the absence of active CNS disease at the time of study entry (screening)
* Patients with a known concurrent malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or carcinoma in situ of the cervix
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2026-07-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Gojo, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (7):
- United States (7):
  - Yale University, New Haven, Connecticut
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level A1: Blinatumomab continuous IV Days 1-28 with Nivolumab 240 mg IV every 2 weeks.
- Dose Level B1: Blinatumomab continuous IV Days 1-28 with Nivolumab 240 mg IV every 2 weeks and Ipilimumab 1 mg/kg IV every 6 weeks.
- Dose Level B-1: Blinatumomab continuous IV Days 1-28 with Nivolumab 80 mg IV every 2 weeks and Ipilimumab 1 mg/kg IV every 6 weeks.
- Dose Expansion (Dose Level A1): Blinatumomab continuous IV Days 1-28 with Nivolumab 80 mg IV every 2 weeks.
Period: Overall Study
Arm/Group | Dose Level A1 | Dose Level B1 | Dose Level B-1 | Dose Expansion (Dose Level A1)
Started | 8 | 3 | 11 | 6
Completed | 6 | 3 | 8 | 6
Not Completed | 2 | 0 | 3 | 0
Not completed — Did not start study treatment | 2 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level A1 | Dose Level B1 | Dose Level B-1 | Dose Expansion (Dose Level A1) | Total
Number analyzed (Participants) | 8 | 3 | 11 | 6 | 28
Age, Continuous [Median (Full Range); unit: Years] | 55 [25 to 75] | 57 [27 to 70] | 54 [33 to 77] | 45 [23 to 84] | 55 [23 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 7 | 2 | 14
  Male | 4 | 2 | 4 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 3 | 9 | 5 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 8 | 3 | 8 | 3 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 11 | 6 | 28
Height [Median (Full Range); unit: centimeter (cm)] | 171.3 [160.0 to 193.0] | 177.8 [174.2 to 181.6] | 167.6 [155.0 to 179.0] | 162.7 [156.5 to 195.0] | 169.5 [155.0 to 195.0]
Weight [Median (Full Range); unit: kilogram (kg)] | 85.5 [71.5 to 100.5] | 96.5 [83.9 to 103.4] | 75.3 [53.4 to 149.7] | 73.4 [66.3 to 103.2] | 83.7 [53.4 to 149.7]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Grade 3, 4, or 5 Adverse Events
Description: Defined by Common Terminology Criteria for Adverse Events, version 5.0. The highest grade experienced by the participant will be reported.
Time Frame: Up to 5.5 years
Population: All participants who started treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A1 | Dose Level B1 | Dose Level B-1 | Dose Expansion (Dose Level A1)
Number analyzed (Participants) | 8 | 3 | 11 | 6
Participants
  Grade 5 | 0 | 1 | 1 | 0
  Grade 4 | 7 | 2 | 7 | 3
  Grade 3 | 1 | 0 | 2 | 2
  Grades 1-2 | 0 | 0 | 1 | 1

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Maximum tolerated dose was determined by the absence of dose limiting toxicity in each patient assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Dose Limiting Toxicities were evaluated during treatment; therefore, the time frame is from the first participant starting treatment to the last participant completing treatment.
Time Frame: Up to 5.5 years
Population: Only participants who started Nivolumab, with or without Ipilimumab, were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A1 | Dose Level B1 | Dose Level B-1 | Dose Expansion (Dose Level A1)
Number analyzed (Participants) | 6 | 3 | 8 | 6
Participants
  Experienced a Dose Limiting Toxicity | 1 | 2 | 1 | 0
  Did not experience a Dose Limiting Toxicity | 5 | 1 | 7 | 6

3. Secondary Outcome: Count of Participants Responders With Minimal Residual Disease
Description: Will be assessed by flow cytometry. Participants who have a clinical response (responders) were evaluated for minimal residual disease negative versus minimal residual disease positive. These are the participants with remission as provided in the Secondary Outcome #4.
Time Frame: Up to 5.5 years
Population: Only participants with a clinical response (i.e. achieving remission) were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A1 | Dose Level B1 | Dose Level B-1 | Dose Expansion (Dose Level A1)
Number analyzed (Participants) | 5 | 3 | 5 | 4
Participants
  Negative MRD | 4 | 3 | 4 | 4
  Positive MRD | 1 | 0 | 1 | 0

4. Secondary Outcome: Number of Participants Achieving Remission
Description: Remission includes participants achieving complete remission or complete remission with incomplete blood count recovery by standard leukemia outcome measures.
Time Frame: Up to 5.5 years
Population: All participants who started treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A1 | Dose Level B1 | Dose Level B-1 | Dose Expansion (Dose Level A1)
Number analyzed (Participants) | 8 | 3 | 11 | 6
Participants
  Achieved remission | 5 | 3 | 5 | 4
  Did not achieve remission | 3 | 0 | 6 | 2

5. Secondary Outcome: Duration of Response
Description: Will be analyzed using the Kaplan Meier method. A sensitivity analysis may be performed to evaluate duration of response while excluding patients who go on to have an allogeneic-hematopoietic stem cell transplantation. Time from measured response to progressive disease, death, or study end, assessed up to 2 years after treatment
Time Frame: Up to 5.5 years
Population: Only responders were included in the analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Dose Level A1 | Dose Level B1 | Dose Level B-1 | Dose Expansion (Dose Level A1)
Number analyzed (Participants) | 5 | 3 | 5 | 4
Days | 205 [116 to 844] | 51 [44 to 828] | 695 [54 to 849] | 490 [155 to 996]

6. Secondary Outcome: Overall Survival
Description: Determined from the first day of treatment on the study until death or last known follow up, assessed up to 2 years after completing treatment.
Time Frame: Up to 5.5 years
Population: Only participants who started nivolumab, with or without ipilimumab, were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Dose Level A1 | Dose Level B1 | Dose Level B-1 | Dose Expansion (Dose Level A1)
Number analyzed (Participants) | 6 | 3 | 8 | 6
Days | 462 [92 to 876] | 182 [86 to 864] | 552 [22 to 910] | 381 [85 to 857]

7. Other Pre Specified Outcome: Changes in Absolute Lymphocyte Count
Description: To examine changes in absolute lymphocyte count before and after blinatumomab and immune checkpoint inhibitor(s) therapy in both peripheral blood and the bone marrow microenvironment. Timeframe is based on duration of treatment.
Time Frame: About 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Distribution of T Cell Subsets and Differentiation Status, Natural Killer (NK) Cells, and B Cells
Description: Will be assessed by flow cytometry. The analyses of pre- and post-treatment peripheral blood and bone marrow specimens for immune parameters will be descriptive and graphical in nature. Data will be summarized for each patient group separately. Flow values at each time point will be summarized using geometric means and standard deviation. Differences in baseline values between patient subgroups will be explored using linear regression models. Timeframe based on duration of treatment.
Time Frame: About 1 year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes in T Cell Co-signaling Receptors Expression
Description: To explore changes in T cell co-signaling receptors expression in defined T cell subpopulations and their canonic transcription factor expression in both peripheral blood and bone marrow before and post-blinatumomab, and immune checkpoint inhibitor(s) therapy. Time frame based on duration of treatment.
Time Frame: About 1 year
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Expression of Co-signaling Molecules on Leukemia Blasts
Description: To examine changes in expression of co-signaling molecules on leukemia blasts (CD10+/CD19+/CD34+) before and after treatment with blinatumomab and checkpoint inhibitors. Time frame based on the duration of treatment.
Time Frame: About 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in Cytokines Levels in Serum
Description: To examine the serum levels of cytokines before and after treatment with blinatumomab and checkpoint inhibitors, including the levels of sCTLA-4. Time frame based on duration of treatment.
Time Frame: About 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Characterization of T Cell Transcriptional Signature
Description: To perform immune profiling of T cell repertoire and characterize T cell transcriptional signature before and after treatment. Time frame based on duration of treatment.
Time Frame: About 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 6.5 years.
Arm/Group | Dose Level A1 | Dose Level B1 | Dose Level B-1 | Dose Expansion (Dose Level A1)
All-Cause Mortality (participants affected / at risk) | 5/8 | 2/3 | 5/11 | 2/6
Serious Adverse Events (participants affected / at risk) | 5/8 | 2/3 | 7/11 | 2/6
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 10/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level A1 (N=8) | Dose Level B1 (N=3) | Dose Level B-1 (N=11) | Dose Expansion (Dose Level A1) (N=6)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Disease Progression (General disorders) | 0 | 0 | 1 | 0
Infusion Related Reaction (General disorders) | 1 | 0 | 0 | 0
Non Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
GVHD (Immune system disorders) | 0 | 1 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 2 | 1
Blood Bilirubin Increased (Investigations) | 1 | 0 | 0 | 1
Platelet Count Decreased (Investigations) | 1 | 0 | 0 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebellar Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient Ischemic Attacks (Nervous system disorders) | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Thromboembolic Event (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level A1 (N=8) | Dose Level B1 (N=3) | Dose Level B-1 (N=11) | Dose Expansion (Dose Level A1) (N=6)
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 5 | 2
Bicarbonate Decrease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Blood Bicarbonate Decreased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Blood LDH Increase (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bone Marrow Hypocellular (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1
Elevated D-dimer (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Elevated Ferritin (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Elevated Fibrinogen (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Elevated Pro-BNP (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 6 | 2
Hyperphosphatemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphocyte Count Increase (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
PT Increased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 2 | 2 | 1
Sinus Tachycardia (Cardiac disorders) | 4 | 1 | 5 | 2
Sinus Trachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 0 | 2 | 0
Blurred Vision (Eye disorders) | 1 | 0 | 1 | 0
Conjunctival Cyst, OS (Eye disorders) | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0 | 1
Floaters (Eye disorders) | 1 | 0 | 1 | 0
Scleral Disorder (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Bloating (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 3 | 2
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 3 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gingival Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Mucositis Oral (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 5 | 1
Oral Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Chills (General disorders) | 3 | 1 | 2 | 3
Edema Face (General disorders) | 0 | 0 | 2 | 0
Edema Limbs (General disorders) | 3 | 0 | 2 | 2
Erythema At PICC Site (General disorders) | 1 | 0 | 0 | 0
Erythema On Scalp (General disorders) | 1 | 0 | 0 | 0
Erythematous Ulcer On Right Upper Pallet (General disorders) | 1 | 0 | 0 | 0
Excoriation Of Buttocks (General disorders) | 1 | 0 | 0 | 0
Excoriation Of Scrotum (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 5 | 3
Fever (General disorders) | 3 | 1 | 5 | 2
Flu Like Symptoms (General disorders) | 1 | 0 | 0 | 0
Gait Disturbance (General disorders) | 1 | 0 | 0 | 0
Infusion Related Reaction (General disorders) | 0 | 0 | 2 | 0
Intermittent PICC Site Irritation (General disorders) | 1 | 0 | 0 | 0
Intermittent PICCsite Irritation (General disorders) | 1 | 0 | 0 | 0
Left Sided Head Numbness (General disorders) | 1 | 0 | 0 | 0
Localized Edema (General disorders) | 0 | 0 | 1 | 0
Non-cardiac Chest Pain (General disorders) | 3 | 0 | 0 | 0
Pain (General disorders) | 4 | 0 | 1 | 0
PICC Site Irritation (General disorders) | 1 | 0 | 0 | 0
Progression Of Disease (General disorders) | 0 | 0 | 1 | 0
Pulmonary Nodules (General disorders) | 1 | 0 | 0 | 0
Rigors (General disorders) | 1 | 0 | 0 | 0
Cytokine Release Syndrome (Immune system disorders) | 2 | 1 | 2 | 4
Hypoimmunoglobulinemia (Immune system disorders) | 0 | 0 | 1 | 0
Bone Infection (Infections and infestations) | 0 | 0 | 0 | 1
Catheter Infection (Infections and infestations) | 1 | 0 | 0 | 0
COVID SARS 2 (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis Infectious (Infections and infestations) | 0 | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 2 | 1
PICC Site Infection (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Viremia (Infections and infestations) | 0 | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hepatotoxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Perianal Lesions (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Postoperative Hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tracheal Hemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 0 | 3 | 0
Alanine Aminotransferase Increased (Investigations) | 4 | 2 | 6 | 2
Alkaline Phosphatase Increased (Investigations) | 4 | 1 | 2 | 0
Aspartate Aminotransferase Increased (Investigations) | 4 | 0 | 6 | 2
Blood Bilirubin Increased (Investigations) | 5 | 0 | 6 | 1
Creatinine Increased (Investigations) | 1 | 0 | 2 | 0
D-Dimer Increase (Investigations) | 0 | 0 | 1 | 0
Fibrinogen Decreased (Investigations) | 1 | 0 | 2 | 0
Generalized Edema (Investigations) | 0 | 0 | 1 | 0
GGT Increased (Investigations) | 1 | 0 | 0 | 0
Hyperphosphatemia (Investigations) | 0 | 0 | 2 | 0
Immunoglobulins Decreased (Investigations) | 0 | 0 | 1 | 0
INR Increased (Investigations) | 0 | 0 | 6 | 0
LDH Increased (Investigations) | 0 | 0 | 1 | 0
Lipase Increased (Investigations) | 3 | 0 | 1 | 1
Lymphocyte Count Decreased (Investigations) | 4 | 2 | 9 | 2
Neutrophil Count Decreased (Investigations) | 4 | 2 | 5 | 3
Platelet Count Decreased (Investigations) | 5 | 2 | 8 | 2
PT Prolonged (Investigations) | 0 | 0 | 1 | 0
Serum Amylase Increased (Investigations) | 1 | 0 | 0 | 0
Weight Gain (Investigations) | 0 | 0 | 2 | 1
Weight Loss (Investigations) | 0 | 1 | 1 | 0
White Blood Cell Decreased (Investigations) | 3 | 2 | 8 | 3
White Blood Cell Increased (Investigations) | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 0
Blood Bicarbonate Decrease (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Glucose Intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 6 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2 | 5 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 4 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1 | 5 | 2
Thiamine Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Zinc Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Bone Infection (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Scattered Pea Size Nodules Bilateral Calfs (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1
Depressed Level Of Consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 4 | 1 | 6 | 3
Memory Impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Movements Involuntary (Nervous system disorders) | 0 | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 2 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1
Sinus Pain (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 4 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 1 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Penile Bleeding (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Tract Pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Genital Edema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatic Obstruction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema RLE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 4 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Excision Of Presumptive Osteomyelitis (Surgical and medical procedures) | 0 | 0 | 0 | 1
Foot Incision And Debridement (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 5 | 2
Hypotension (Vascular disorders) | 1 | 0 | 3 | 0
Non-occlusive Thrombus (Vascular disorders) | 0 | 0 | 1 | 0
Superficial Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT02879695/Prot_SAP_000.pdf